CLINICAL TRIAL: NCT02379949
Title: Virtual Reality Exposure Therapy for the Treatment of Social Phobia
Acronym: FOPSII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Virtually Better, Inc. (Industry)
Responsible Party: Principal Investigator, Page Anderson, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R42MH060506-02 (NIH)
Record Dates: First submitted 2015-01-29; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Social Anxiety Disorder
Keywords: virtual reality exposure therapy; social phobia; social anxiety disorder; cognitive behavioral therapy
MeSH Terms: conditions — Phobia, Social | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Virtual Reality Exposure Therapy (Experimental): During virtual reality exposure therapy, a person encounters a feared stimulus (public speaking) in a computer-generated environment.
  Interventions: Behavioral: Virtual Reality Exposure Therapy
- Exposure Group Therapy (Active Comparator): Exposure Group Therapy a behavioral treatment for social phobia. Participants face their fears by giving speeches to other group members.
  Interventions: Behavioral: Exposure Group Therapy
- Waitlist (No Intervention): Participants assigned to wait list were re-randomized to virtual reality exposure therapy or exposure group therapy following the waiting period.

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy — During virtual reality exposure therapy, a person encounters a feared stimulus (public speaking) in a computer-generated environment.
  Arms: Virtual Reality Exposure Therapy
Behavioral: Exposure Group Therapy — Exposure Group Therapy a behavioral treatment for social phobia. Participants face their fears by giving speeches to other group members.
  Arms: Exposure Group Therapy

SUMMARY:
This randomized clinical trial compares virtual reality exposure therapy to exposure group therapy to a waiting list control group.

DETAILED DESCRIPTION:
Virtual reality exposure therapy (VRE) for the treatment of anxiety disorders has received considerable attention. During VRE, a person encounters a feared stimulus in a computer-generated environment, often through the use of a head mounted display and motion tracker that allows for multisensory input and natural movement. Several advantages of VRE have been noted - both clinical, such as treatment acceptability, and methodological, such as the ability to conduct exposure in a tightly controlled environment. Empirical support for VRE varies across anxiety disorders. Specifically, randomized controlled trials support the efficacy of VRE with fear of flying and acrophobia and show that it is equally effective as in vivo exposure. These phobias lend themselves well to VRE; the feared stimulus is circumscribed and contains powerful physical cues that can be produced within a virtual environment. There is less controlled research on the use of VRE for other anxiety disorders. The current study examines VRE for social anxiety disorder, which is characterized by fear of negative evaluation, and thus may be more difficult to evoke and treat using a virtual environment. Further, no research to date has compared VRE and the gold standard treatment for social anxiety disorder - cognitive behavioral therapy in a group format.

The purpose of the current study is to compare VRE and Exposure Group Therapy to wait list in a sample of adults meeting criteria for social anxiety disorder with a primary fear of public speaking. It is hypothesized that, relative to wait list, those receiving treatment will improve on standardized measures of public speaking fears and fears of negative evaluation, as well as a behavioral avoidance task. Participants also are expected to maintain treatment gains at 3 and 12-month follow-up. Comparisons between the two active treatments also will be made.

Procedure

Following consent, study candidates completed a phone interview to screen for obvious exclusion criteria (e.g., current treatment for social anxiety disorder) and then an in-person, pretreatment assessment consisting of the Structured Clinical Interview for the DSM-IV (SCID), speech task, and the battery of self-report measures. Eligible participants were randomly assigned to virtual reality exposure therapy, exposure group therapy, or wait list by simple randomization using a computerized random number generator. Concealment procedures were used to prevent foreknowledge of treatment assignment from influencing enrollment. Each potential participant had a participant number, which was only known by the study coordinator. The first author kept a hard copy of a list linking participant number to condition assignment in a locked file drawer. Once a participant was enrolled, the study coordinator asked for the treatment condition for a particular participant number. The first author had no knowledge of which participant was linked with a participant number, and the study coordinator had no knowledge of which participant number was linked with treatment condition. Participants assigned to wait list were re-randomized to virtual reality exposure therapy or exposure group therapy following the waiting period (Figure 1). Participants completed all assessment and treatment sessions at a psychology clinic within at an urban research university that is accessible by public transportation.

Assessments

Participants completed assessments at pretreatment, posttreatment, and follow-up. Self-report outcome measures were completed at each assessment point. Participants were asked to complete the behavioral avoidance task at pretreatment and posttreatment. The anxiety, mood, and substance use modules of the SCID were administered at pretreatment, and the anxiety module was administered at the 3-month follow-up.

All assessments were conducted by doctoral students who were blind to the type of treatment to be received. All pretreatment and follow-up diagnostic assessments were videotaped, and a randomly selected subset (N=10) were reviewed by a licensed psychologist to calculate the inter-rater reliability of pretreatment assessment (100% agreement for primary diagnosis, with one disagreement on severity). Compensation was provided to participants who completed the self-report battery of measures administered at posttreatment, 3- and 12-month follow-up.

Treatment

Prior to administering therapy, study therapists attended two day training workshops for each treatment, led by the developers of the respective treatments. Each study therapist also received weekly supervision by the first author. There were 5 study therapists: 2 licensed clinical psychologists with experience in manualized treatment, and 3 doctoral students with no experience with manualized treatments. All therapists administered both treatments.

Both treatments were administered according to a manualized protocol for 8 sessions. The VRE and EGT treatment groups were designed to be as similar as possible, with the exception of the modality for the delivery of exposure. Both treatments began with a treatment rationale and psychoeducation about social anxiety disorder. During sessions 2- 8, both treatments addressed specific aspects of social anxiety disorder identified in psychopathology literature, including self-focused attention, perceptions of self and others, perceptions of emotional control, rumination, realistic goal setting for social situations through the use of such techniques as cognitive preparation, and challenging of cost and probability biases. Session 8 also included relapse prevention. Homework was assigned for both treatments, including a daily mirror task, daily record of social situations, and identification of cognitive biases.

Virtual Reality Exposure (VRE)

Virtual environments included a virtual conference room (~5 audience members), a virtual classroom (~35 audience members), and a virtual auditorium (100+ audience members). Therapists could manipulate audience reactions in a number of ways including making them appear interested, bored, supportive, hostile, distracted (i.e., cell phone ringing). Virtual audience members could also pose questions, either standardized (e.g., "I don't understand, could you explain again") or tailored to the client using therapist voice-over. Virtual environments were manipulated according to the participants fear hierarchy. Participants were exposed to each item on their hierarchy until their fear decreased.

Exposure Group Therapy (EGT)

EGT was co-led by a licensed clinical psychologist and an advanced doctoral student. Groups consisted of up to five participants. During exposure, participants gave a videotaped speech in front of the group. Group members were also asked to provide each other with positive feedback when the videotaped speeches were reviewed.

Every effort was made to equate time in exposure across treatment group. Participants receiving VRE completed 4 trials of exposure. Because of the risk of simulator sickness (e.g., headaches, nausea), exposure trials lasted no longer than 30 minutes, for a total of up to 120 minutes. Participants receiving EGT received 6 trials of exposure. The amount of time spent on each group member varied according to the number of participants in the group. On average, for a group with 4 participants, participants completed 6 trials of exposure for 20 minutes for a total of 120 minutes.

Wait List

After 8 weeks, wait list participants completed the self-report battery. Wait list participants were re-randomized to either virtual reality exposure or exposure group therapy following the waiting period and received the same 8-week treatment protocol described above.

ELIGIBILITY:
Inclusion Criteria:

* Speakers of English meeting DSM-IV (APA, 2000) criteria for a primary diagnosis of social anxiety disorder
* Self-identifying public speaking as their primary social fear
* Participants were required to be stabilized on psychoactive medication(s) and dosage(s) for 3 months.

Exclusion Criteria:

* history of mania, schizophrenia, or psychosis
* current suicidal ideation, alcohol, or substance dependence
* inability to tolerate the virtual reality helmet/environment
* history of seizures
* concurrent psychotherapy for social anxiety disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2004-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Personal Report of Confidence as a Speaker | Post-treatment, approximately 8 weeks after initial screening session
  30 true/false items measuring public speaking confidence across three dimensions: before, during, and after delivering a speech.
Fear of Negative Evaluation-Brief Form | Post-treatment, approximately 8 weeks after initial screening session
  12-item questionnaire measuring the degree to which individuals fear being negatively evaluated by others across a number of social settings.
Behavioral Avoidance Test | Post-treatment, approximately 8 weeks after initial screening session
  The behavioral avoidance test was based on a standardized speech assessment protocol (Beidel, Turner, Jacob, & Cooley, 1989), in which participants are given 3 min to prepare notes on five controversial topics (e.g., abortion, same-sex marriage). Participants are then asked to speak for 10 min on up to three topics and to rate how well they performed (0 -10) and how anxious they felt (0 -10), with higher numbers indicating better performance and higher anxiety. Audience members consisted of two to four trained undergraduate or graduate students; the therapist was never an audience member
Clinician Global Impressions of Improvement | Post-treatment, approximately 8 weeks after initial screening session
  A clinician-rated, global measure of change in severity of symptoms, ranging from 1 (very much improved) to 7 (very much worse).
Personal Report of Confidence as a Speaker | 3 months following final treatment session
  30 true/false items measuring public speaking confidence across three dimensions: before, during, and after delivering a speech.
Fear of Negative Evaluation-Brief Form | 3 months following final treatment session
  30 true/false items measuring public speaking confidence across three dimensions: before, during, and after delivering a speech.
Behavioral Avoidance Test | 3 months following final treatment session
  The behavioral avoidance test was based on a standardized speech assessment protocol (Beidel, Turner, Jacob, & Cooley, 1989), in which participants are given 3 min to prepare notes on five controversial topics (e.g., abortion, same-sex marriage). Participants are then asked to speak for 10 min on up to three topics and to rate how well they performed (0 -10) and how anxious they felt (0 -10), with higher numbers indicating better performance and higher anxiety. Audience members consisted of two to four trained undergraduate or graduate students; the therapist was never an audience member
Clinician Global Impressions of Improvement | 3 months following final treatment session
  A clinician-rated, global measure of change in severity of symptoms, ranging from 1 (very much improved) to 7 (very much worse).
Personal Report of Confidence as a Speaker | 12 months following final treatment session
  30 true/false items measuring public speaking confidence across three dimensions: before, during, and after delivering a speech.
Fear of Negative Evaluation-Brief Form | 12 months following final treatment session
  12-item questionnaire measuring the degree to which individuals fear being negatively evaluated by others across a number of social settings.
Behavioral Avoidance Test | 12 months following final treatment session
  The behavioral avoidance test was based on a standardized speech assessment protocol (Beidel, Turner, Jacob, & Cooley, 1989), in which participants are given 3 min to prepare notes on five controversial topics (e.g., abortion, same-sex marriage). Participants are then asked to speak for 10 min on up to three topics and to rate how well they performed (0 -10) and how anxious they felt (0 -10), with higher numbers indicating better performance and higher anxiety. Audience members consisted of two to four trained undergraduate or graduate students; the therapist was never an audience member.
Clinician Global Impressions of Improvement | 12 months following final treatment session
  The behavioral avoidance test was based on a standardized speech assessment protocol (Beidel, Turner, Jacob, & Cooley, 1989), in which participants are given 3 min to prepare notes on five controversial topics (e.g., abortion, same-sex marriage). Participants are then asked to speak for 10 min on up to three topics and to rate how well they performed (0 -10) and how anxious they felt (0 -10), with higher numbers indicating better performance and higher anxiety. Audience members consisted of two to four trained undergraduate or graduate students; the therapist was never an audience member.

CONTACTS AND LOCATIONS:
Overall Officials: Page L Anderson, Ph.D., Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Anderson PL, Zimand E, Hodges LF, Rothbaum BO. Cognitive behavioral therapy for public-speaking anxiety using virtual reality for exposure. Depress Anxiety. 2005;22(3):156-8. doi: 10.1002/da.20090. PMID 16231290
- [Background] Anderson, P., Rothbaum, B. O., & Hodges, L. F. Virtual reality exposure in the treatment of social anxiety. Cognitive and Behavioral Practice, 10: 240-247, 2003.
- [Background] Andersson G, Carlbring P, Holmstrom A, Sparthan E, Furmark T, Nilsson-Ihrfelt E, Buhrman M, Ekselius L. Internet-based self-help with therapist feedback and in vivo group exposure for social phobia: a randomized controlled trial. J Consult Clin Psychol. 2006 Aug;74(4):677-86. doi: 10.1037/0022-006X.74.4.677. PMID 16881775
- [Background] APA. Diagnostic and statistical manual of mental disorders, Fourth Edition - Text Revision (4th ed.): American Psychiatric Publishing, Inc. 2000.
- [Background] Attkisson, C.C. & Greenfield, T.K.The UCSF client satisfaction scales: I. The Client Satisfaction Questionnaire-8. In M.E. Maruish (Ed.), The use of psychological testing for treatment planning and outcomes assessment (2nd ed., pp. 1333-1346). Mahwah, NJ: Erlbaum. 1999.
- [Background] Beck, A. T., Steer, R. A., & Brown, G. K. (1996). Manual for Beck Depression Inventory - II. San Antonio, TX: The Psychological Corporation, Harcourt, Brace & Company.
- [Background] Beidel, D. C., Turner, S. M., Jacob, R. G., & Cooley, M. R. Assessment of social phobia: Reliability of an impromptu speech task. Journal of Anxiety Disorders, 3: 149-158, 1989.
- [Background] Blote AW, Kint MJ, Miers AC, Westenberg PM. The relation between public speaking anxiety and social anxiety: a review. J Anxiety Disord. 2009 Apr;23(3):305-13. doi: 10.1016/j.janxdis.2008.11.007. Epub 2008 Nov 25. PMID 19117721
- [Background] Borkovec, T. D., & Nau, S. D. Credibility of analogue therapy rationales. Journal of Behavior Therapy and Experimental Psychiatry, 3: 257- 260, 1972.
- [Background] Botella, C., Gallego, M. J., Garcia-Palacios, A., Baños, R. M., Quero, S., & Guillen, V. An internet-based self-help program for the treatment of fear of public speaking: A case study. Journal of Technology in Human Services, 26: 182-202, 2008.
- [Background] Botella, C., García-Palacios, A., Villa, H., Baños, R. M., Quero, S., Alcañiz, M., & Riva, G. Virtual reality exposure in the treatment of panic disorder and agoraphobia: A controlled study. Clinical Psychology & Psychotherapy, 14: 164-175, 2007.
- [Background] Bouchard, S., Dumoulin, S., Robillard, G., Guitard, T. & Klinger, E. et al. A randomized control trial for the use of in virtuo exposure in the treatment of social phobia: final results. Journal of CyberTherapy and Rehabilitation, 4: 197-199, 2011.
- [Background] Bouton, M. E., Woods, A. M., Moody, E. W., Sunsay, C., & Garcia-Guitierrez, A. (2006). Counteracting the context-dependence of extinction: Relapse and some tests of possible methods of relapse prevention. In M. G. Craske, D. Hermans, & D. Vansteenwegen (Eds.), Fear and learning: Basic science to clinical application. (pp.175-196). Washington, DC: American Psychological Association.
- [Background] Busseri MA, Tyler JD. Interchangeability of the Working Alliance Inventory and Working Alliance Inventory, Short Form. Psychol Assess. 2003 Jun;15(2):193-7. doi: 10.1037/1040-3590.15.2.193. PMID 12847779
- [Background] Collins KA, Westra HA, Dozois DJ, Stewart SH. The validity of the brief version of the Fear of Negative Evaluation Scale. J Anxiety Disord. 2005;19(3):345-59. doi: 10.1016/j.janxdis.2004.02.003. PMID 15686861
- [Background] Clark, D. M., & Wells, A. (1995). A cognitive model of social phobia. In R. G. Heimberg, M. R. Liebowitz, D. A. Hope, & F. R. Schneier (Eds.), Social phobia: Diagnosis, assessment, and treatment (pp. 69-93). New York: Guilford Press.
- [Background] Emmelkamp PM. Technological innovations in clinical assessment and psychotherapy. Psychother Psychosom. 2005;74(6):336-43. doi: 10.1159/000087780. PMID 16244509
- [Background] Emmelkamp PM, Krijn M, Hulsbosch AM, de Vries S, Schuemie MJ, van der Mast CA. Virtual reality treatment versus exposure in vivo: a comparative evaluation in acrophobia. Behav Res Ther. 2002 May;40(5):509-16. doi: 10.1016/s0005-7967(01)00023-7. PMID 12038644
- [Background] Feingold A. Effect sizes for growth-modeling analysis for controlled clinical trials in the same metric as for classical analysis. Psychol Methods. 2009 Mar;14(1):43-53. doi: 10.1037/a0014699. PMID 19271847
- [Background] First, M. B., Spitzer, R. L., Gibbon, M., & Williams, J. B. W. (1994). Structured Clinical Interview for Axis I DSM-IV Disorders-Research Edition. New York, NY: Biometrics Research Department.
- [Background] Fresco DM, Coles ME, Heimberg RG, Liebowitz MR, Hami S, Stein MB, Goetz D. The Liebowitz Social Anxiety Scale: a comparison of the psychometric properties of self-report and clinician-administered formats. Psychol Med. 2001 Aug;31(6):1025-35. doi: 10.1017/s0033291701004056. PMID 11513370
- [Background] Guy, W. (1976) ECDEU Assessment Manual for Psychotherapy - Revised (DHEW Publication No. ADM 76-338). Bethesda, MD: National Institute of Mental Health.
- [Background] Hofmann SG. Cognitive mediation of treatment change in social phobia. J Consult Clin Psychol. 2004 Jun;72(3):392-399. doi: 10.1037/0022-006X.72.3.392. PMID 15279523
- [Background] Hofmann SG. Cognitive factors that maintain social anxiety disorder: a comprehensive model and its treatment implications. Cogn Behav Ther. 2007;36(4):193-209. doi: 10.1080/16506070701421313. PMID 18049945
- [Background] Hofmann SG, Dibartolo PM. An instrument to assess self-statements during public speaking: scale development and preliminary psychometric properties. Behav Ther. 2000;31(3):499-515. doi: 10.1016/s0005-7894(00)80027-1. PMID 16763666
- [Background] Horvath, A. O., & Greenberg, L. S. Development and validation of the Working Alliance Inventory. Journal of Counseling Psychology, 36: 223-233, 1989.
- [Background] Klinger E, Bouchard S, Legeron P, Roy S, Lauer F, Chemin I, Nugues P. Virtual reality therapy versus cognitive behavior therapy for social phobia: a preliminary controlled study. Cyberpsychol Behav. 2005 Feb;8(1):76-88. doi: 10.1089/cpb.2005.8.76. PMID 15738695
- [Background] Klorman, R., Weerts, T. C., Hastings, J. E., Melamed, B. G., & Lang, P. J. Psychometric description of some specific-fear questionnaires. Behavior Therapy, 5: 401-409, 1974.
- [Background] Leary, M. R. A brief version of the Fear of Negative Evaluation Scale. Personality and Social Psychology Bulletin, 9: 371- 375, 1983.
- [Background] McCroskey, J. C. Validity of the PRCA as an index of oral communication apprehension. Communication Monographs, 45: 192-203, 1978.
- [Background] McGilloway S, Mhaille GN, Bywater T, Furlong M, Leckey Y, Kelly P, Comiskey C, Donnelly M. A parenting intervention for childhood behavioral problems: a randomized controlled trial in disadvantaged community-based settings. J Consult Clin Psychol. 2012 Feb;80(1):116-127. doi: 10.1037/a0026304. Epub 2011 Dec 12. PMID 22148879
- [Background] Meyerbroker K, Emmelkamp PM. Virtual reality exposure therapy in anxiety disorders: a systematic review of process-and-outcome studies. Depress Anxiety. 2010 Oct;27(10):933-44. doi: 10.1002/da.20734. PMID 20734361
- [Background] Meyerbroker, K., & Emmelkamp, P. M. G. Therapeutic processes in virtual reality exposure therapy: The role of cognitions and the therapeutic alliance. Journal of Cyber Therapy and Rehabilitation, 1: 247-257, 2008.
- [Background] Muthén, L. K., & Muthén, B. O. (2012). Mplus user's guide (6th ed.). Los Angeles, CA: Muthén & Muthén.
- [Background] Opris D, Pintea S, Garcia-Palacios A, Botella C, Szamoskozi S, David D. Virtual reality exposure therapy in anxiety disorders: a quantitative meta-analysis. Depress Anxiety. 2012 Feb;29(2):85-93. doi: 10.1002/da.20910. Epub 2011 Nov 7. PMID 22065564
- [Background] Otto, M. W., Smits, J. A. J., & Reese, H. E. Combined psychotherapy and pharmacotherapy for mood and anxiety disorders in adults: Review and analysis. Clinical Psychology: Science and Practice, 12: 72-86, 2005.
- [Background] Parsons TD, Rizzo AA. Affective outcomes of virtual reality exposure therapy for anxiety and specific phobias: a meta-analysis. J Behav Ther Exp Psychiatry. 2008 Sep;39(3):250-61. doi: 10.1016/j.jbtep.2007.07.007. Epub 2007 Jul 25. PMID 17720136
- [Background] Paul, G. L. (1966). Insight vs desensitization in psychotherapy. Standford, CA: Stanford University Press.
- [Background] Piaggio G, Elbourne DR, Altman DG, Pocock SJ, Evans SJ; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: an extension of the CONSORT statement. JAMA. 2006 Mar 8;295(10):1152-60. doi: 10.1001/jama.295.10.1152. PMID 16522836
- [Background] Phillips GC, Jones GE, Rieger ER, Snell JB. Normative data for the personal report of confidence as a speaker. J Anxiety Disord. 1997 Mar-Apr;11(2):215-20. doi: 10.1016/s0887-6185(97)00007-8. PMID 9168343
- [Background] Powers MB, Emmelkamp PM. Virtual reality exposure therapy for anxiety disorders: A meta-analysis. J Anxiety Disord. 2008;22(3):561-9. doi: 10.1016/j.janxdis.2007.04.006. Epub 2007 Apr 27. PMID 17544252
- [Background] Rapee RM, Gaston JE, Abbott MJ. Testing the efficacy of theoretically derived improvements in the treatment of social phobia. J Consult Clin Psychol. 2009 Apr;77(2):317-27. doi: 10.1037/a0014800. PMID 19309190
- [Background] Raudenbush, S.W. and Bryk, A.S. (2002). Hierarchical Linear Models (Second Edition). Thousand Oaks: Sage Publications.
- [Background] Raudenbush SW, Xiao-Feng L. Effects of study duration, frequency of observation, and sample size on power in studies of group differences in polynomial change. Psychol Methods. 2001 Dec;6(4):387-401. PMID 11778679
- [Background] Rothbaum BO, Hodges L, Smith S, Lee JH, Price L. A controlled study of virtual reality exposure therapy for the fear of flying. J Consult Clin Psychol. 2000 Dec;68(6):1020-6. doi: 10.1037//0022-006x.68.6.1020. PMID 11142535
- [Background] Safir MP, Wallach HS, Bar-Zvi M. Virtual reality cognitive-behavior therapy for public speaking anxiety: one-year follow-up. Behav Modif. 2012 Mar;36(2):235-46. doi: 10.1177/0145445511429999. Epub 2011 Dec 15. PMID 22180390
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):834-40. doi: 10.1016/j.jclinepi.2010.02.005. Epub 2010 Mar 25. No abstract available. PMID 20346629
- [Background] Shiban Y, Pauli P, Muhlberger A. Effect of multiple context exposure on renewal in spider phobia. Behav Res Ther. 2013 Feb;51(2):68-74. doi: 10.1016/j.brat.2012.10.007. Epub 2012 Nov 11. PMID 23261707
- [Background] Taylor CT, Alden LE. Safety behaviors and judgmental biases in social anxiety disorder. Behav Res Ther. 2010 Mar;48(3):226-37. doi: 10.1016/j.brat.2009.11.005. Epub 2009 Nov 18. PMID 19954772
- [Background] Van Breukelen GJ. ANCOVA versus change from baseline: more power in randomized studies, more bias in nonrandomized studies [corrected]. J Clin Epidemiol. 2006 Sep;59(9):920-5. doi: 10.1016/j.jclinepi.2006.02.007. Epub 2006 Jun 23. PMID 16895814
- [Background] Wallach HS, Safir MP, Bar-Zvi M. Virtual reality cognitive behavior therapy for public speaking anxiety: a randomized clinical trial. Behav Modif. 2009 May;33(3):314-38. doi: 10.1177/0145445509331926. Epub 2009 Mar 25. PMID 19321811
- [Background] Whaley AL, Davis KE. Cultural competence and evidence-based practice in mental health services: a complementary perspective. Am Psychol. 2007 Sep;62(6):563-74. doi: 10.1037/0003-066X.62.6.563. PMID 17874897
- [Background] Zaider TI, Heimberg RG, Fresco DM, Schneier FR, Liebowitz MR. Evaluation of the clinical global impression scale among individuals with social anxiety disorder. Psychol Med. 2003 May;33(4):611-22. doi: 10.1017/s0033291703007414. PMID 12785463